CLINICAL TRIAL: NCT03599791
Title: Multicentre, Randomized, Double-blind, Parallel Group Phase III Study to Assess Efficacy and Safety of Dymista® Compared to Azep® and Flixonase® Nasal Sprays in the Treatment of Chinese Patients With Allergic Rhinitis/Rhinoconjunctivitis
Brief Title: DYmista NAsal Spray in CHInese Patients
Acronym: DYNAS-CHI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X-03065-3303
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2020-02

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; hayfever; rhinoconjunctivitis; azelastine; fluticasone; nasal spray; seasonal; perennial; TNSS; TOSS
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — azelastine; Fluticasone

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, double-blind, active controlled, parallel group study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Azelastine Hydrochl. + Fluticasone Prop. (Experimental): Drug: Azelastine Hydrochl./Fluticasone Prop. 0.137/0.05 MG/ACTUAT Nasal Spray, consists of a fixed-dose combination of azelastine hydrochloride and fluticasone propionate; 1 spray per nostril twice daily for 14 days, with 3 to 7 days of lead-in period. At a certain point during the study, patients will receive Placebo.
  Interventions: Drug: Azelastine Hydrochl./Fluticasone Prop. 0.137/0.05 MG/ACTUAT
- Azelastine hydrochloride (Active Comparator): Drug: Azelastine Hydrochloride 0.137 MG/ACTUAT Nasal Spray, 1 spray per nostril twice daily for 14 days, with 3 to 7 days of lead-in period. At a certain point during the study, patients will receive Placebo.
  Interventions: Drug: Azelastine Hydrochloride 0.137 MG/ACTUAT
- Fluticasone propionate (Active Comparator): Drug: Fluticasone Propionate 0.05 MG/ACTUAT Nasal Spray, 1 spray per nostril twice daily for 14 days, with 3 to 7 days of lead-in period. At a certain point during the study, patients will receive Placebo.
  Interventions: Drug: Fluticasone Propionate 0.05 MG/ACTUAT

INTERVENTIONS:
Drug: Azelastine Hydrochl./Fluticasone Prop. 0.137/0.05 MG/ACTUAT — Dymista Nasal spray suspension
  Other Names: Dymista
  Arms: Azelastine Hydrochl. + Fluticasone Prop.
Drug: Azelastine Hydrochloride 0.137 MG/ACTUAT — AZEP Nasal spray solution
  Other Names: AZEP
  Arms: Azelastine hydrochloride
Drug: Fluticasone Propionate 0.05 MG/ACTUAT — Fluticasone propionate nasal spray suspension
  Other Names: Flixonase
  Arms: Fluticasone propionate

SUMMARY:
This study is a phase III clinical study to assess the efficacy and safety of Dymista® Nasal Spray in comparison to Azep® nasal spray and Flixonase® nasal spray in Chinese patients aged ≥ 12 years with moderate-to-severe allergic rhinitis/rhinoconjunctivitis.

DETAILED DESCRIPTION:
This is a multicentre, randomized, active controlled prospective clinical trial in adult and adolescent patients with AR (seasonal and/or perennial), who have moderate-to-severe symptoms (rhinitis/ rhinoconjunctivitis), based on the Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 Guidelines. The study consists of a 3 to 7-day Lead-in Period during which patients must meet a minimum symptom severity score to be eligible for the Treatment Period. All patients will start the Lead-in Period straight after Screening Visit as soon as in/exclusion criteria are fulfilled. The Lead-in Period will be followed by a 14-day double-blind Treatment Period. At some time point during the study, patients will receive Placebo and Dymista® nasal spray or Azep® nasal spray or Flixonase® nasal spray, 1 spray per nostril twice daily according to randomization. On the first day of the Lead-in Period patients must meet study inclusion/exclusion criteria and have a sufficient AR symptom score to qualify for entry. Qualified patients will be requested to keep a Diary of nasal and ocular symptoms throughout the study period. Additionally, patients will be requested to complete the Adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) and EuroQoL 5D questionnaire (EQ-5D) on Day 1, Day 8 and Day 15. Both Questionnaires will be completed by adult patients only.

ELIGIBILITY:
General Inclusion Criteria:

To be eligible for enrolment into this study, a patient must comply with all of the following criteria:

1. Male or female patient 12 years of age or older.
2. Provide written informed consent.
3. Patients must have moderate-to-severe rhinitis or rhinoconjunctivitis, defined as rhinitis/rhinoconjunctivitis with one or more of the following being present:

   * Sleep disturbance.
   * Impairment of daily activities, leisure and/or sport.
   * Impairment of learning or work.
   * Troublesome symptoms.
4. Patients must have moderate-to-severe rhinitis or rhinoconjunctivitis and monotherapy with either intranasal antihistamine or glucocorticoid is not considered sufficient at the discretion of the Investigator and/or designee.
5. Conducting the Lead-in Period according to the protocol.
6. Willing and able to comply with the study requirements.
7. At least a 2-year history of AR (seasonal and/or perennial) during the same time of year as the scheduled study time.
8. The presence of Immunoglobulin E (IgE)-mediated hypersensitivity to one or more aeroallergens present in current patient environment, confirmed by a positive response to an established standard diagnostic test at the site within the last year (before randomization).
9. General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the Investigator or the sponsor's medical officer. When in doubt, the Investigator should confer with the sponsor's medical monitor or designee to determine eligibility for the study.
10. Patient agrees to avoid prohibited medication and alcohol and use effective methods of contraception during the study.
11. Negative pregnancy test in women with childbearing potential.

General Exclusion Criteria:

A patient is ineligible and must not enter the study if any of the following criteria is met:

Safety concerns:

1. Presence of any hypersensitivity to drugs similar to azelastine hydrochloride, fluticasone propionate, or to any of the excipients.
2. Women who are pregnant or nursing.
3. Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception.
4. Clinically significant arrhythmia (or unstable despite medical treatment) or symptomatic cardiac conditions.
5. A known history of alcohol or drug abuse within the last 2 years.
6. Diagnosis of human immunodeficiency virus (HIV) infection.
7. Patients with a diagnosis of Glaucoma, cataract, or central serous chorioretinopathy (CSCR).

   Lack of suitability for the study:
8. Nasal disease(s) likely to affect deposition of intranasal medication, such as sinusitis, rhinitis medicamentosa, clinically significant polyposis, or nasal structural abnormalities (e.g. nasal septum deviation).
9. Nasal surgery or sinus surgery within the previous year.
10. Chronic sinusitis - more than 3 episodes per year.
11. Major malignancies including pheochromocytoma within the last 5 years. Exception will be considered where malignancies have been resolved as judged by Investigator.
12. The use of any investigational drug within 30 days prior to Screening Visit. No other investigational products are permitted for use during the conduct of this study.
13. Respiratory Tract Infections including within 14 days prior to Screening Visit.
14. Asthma (with the exception of mild intermittent asthma). Patients with mild intermittent asthma who only require short-acting inhaled bronchodilators and who do not have nocturnal awakening as a result of asthma are eligible for enrolment.
15. Other significant diseases of bronchus and lungs including chronic obstructive pulmonary disease (COPD), emphysema, bronchiectasis, tuberculosis, pneumonia.
16. Any surgical or medical condition or physical or laboratory findings, which in the opinion of the Investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug; that might significantly affect the patient's ability to complete this trial; or their safety in this trial.
17. Clinically relevant abnormal physical findings during the Lead-in Period which, in the opinion of the Investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures.
18. Current use or expected requirement of ritonavir or strong P4503A4 inhibitors including cobicistat-containing products.
19. Specific immunotherapy within 6 months prior to Screening Visit. If the patient received immunotherapy a 6-month washout period is required following the last dose of immunotherapy.
20. Use of certain medications or therapies (e.g. for Allergic Rhinitis) within a specified time period

    Administrative reasons:
21. Planned travel outside of the aeroallergen area during the study period.
22. Employees of the Sponsor, research centre or private practice and their family members.
23. Start-of-treatment Visit (Day 1): have not fully completed Diary.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Combined 12-hour rTNSS (AM + PM) | 14 days
  Total nasal symptom score (TNSSS) is a sum of 4 individual nasal symptom scores: nasal itching, runny nose, congestion and sneezing. Each nasal symptom will be assessed according to a 4-ponit scale (0 = no, 1 = mild, 2 = moderate, 3 = severe symptom); thus, each TNSS will be in the range from 0 (no symptoms at all) to 12 (all 4 symptoms are severe) and the combined 12-hour reflective TNSS (morning + evening) will be in the range of 0 to 24 accordingly

CONTACTS AND LOCATIONS:
Overall Officials: DucTung Nguyen, Dr., Study Director — Meda Pharma GmbH & Co. KG (A Mylan Company)
Locations (33):
- China (33):
  - Investigational Site 2, Beijing, Beijing Municipality
  - Investigational Site 3, Beijing, Beijing Municipality
  - Investigational Site 4, Beijing, Beijing Municipality
  - Investigational Site 5, Beijing, Beijing Municipality
  - Investigational Site, Chongqing, Chonqing
  - Investigational Site 1, Beijing, Dongcheng District
  - Investigational Site 1, Guangzhou, Guangdong
  - Investigational Site 2, Guangzhou, Guangdong
  - Investigational Site 1, Wuhan, Hubei
  - Investigational Site 2, Wuhan, Hubei
  - Investigational Site, Changsha, Hunan
  - Investigational Site, Nanchang, Jiangxi
  - Investigational Site, Changchun, Jilin
  - Investigational Site, Tonghua, Jilin
  - Investigational Site, Yanbian, Jilin
  - Investigational Site, Jining, Jining
  - Investigational Site, Dalian, Liaoning
  - Investigational Site, Nanjing, Nanjing
  - Investigational Site 1, Qingdao, Shandong
  - Investigational Site 2, Qingdao, Shandong
  - Investigational Site, Yantai, Shangdong
  - Investigational Site, Zibo, Shangdong
  - Investigational Site, Shanghai, Shanghai Municipality
  - Investigational Site, Changzhi, Shanxi
  - Investigational Site, Taiyuan, Shanxi
  - Investigational Site 1, Xi’an, Shanxi
  - Investigational Site 2, Xi’an, Shanxi
  - Investigational Site, Chengdu, Sichuan
  - Investigational Site 1, Tianjin, Tianjin Municipality
  - Investigational Site 2, Tianjin, Tianjin Municipality
  - Investigational Site 3, Tianjin, Tianjin Municipality
  - Investigational Site 4, Tianjin, Tianjin Municipality
  - Investigational Site, Ürümqi, Xianjiang Uygur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou B, Cheng L, Pan J, Wang H, Jin Y, Zhao C, Lin P, Tan G, Fang H, Zhang H, Zhou H, Dong Y, Kuhl HC, Ramalingam RK, Nguyen DT. A Clinical Study to Assess the Efficacy and Safety of MP-AzeFlu Nasal Spray in Comparison to Commercially Available Azelastine Hydrochloride and Fluticasone Propionate Nasal Sprays in Chinese Volunteers with Allergic Rhinitis. Pulm Ther. 2023 Sep;9(3):411-427. doi: 10.1007/s41030-023-00238-8. Epub 2023 Aug 14. PMID 37580498